CLINICAL TRIAL: NCT05166525
Title: Kaiser Permanente Evaluation of Medically-Tailored Meals in Adults With Chronic Medical Conditions at High Readmission Risk (KP NOURISH) Study
Brief Title: Kaiser Permanente Evaluation of Medically Tailored Meals in Adults With Medical Conditions at High Readmission Risk
Acronym: KP NOURISH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1527031
Record Dates: First submitted 2021-12-08; First posted 2021-12-22 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Heart Failure; Chronic Kidney Diseases; Diabetes Mellitus, Type 2
Keywords: Medically Tailored Meals; Nutritional Counseling; Food is Medicine
MeSH Terms: conditions — Heart Failure; Renal Insufficiency, Chronic; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: This study is a virtual, remote, decentralized pragmatic clinical trial comparing the efficacy of medically tailored meals alone or medically tailored meals with remote nutritional counseling compared with usual standard of care in adults with a targeted, nutrition-sensitive chronic medical condition (heart failure, diabetes mellitus, chronic kidney disease)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Medically tailored meals only (Active Comparator): Receive medically-tailored meals only (1 meal per day for total of 10 weeks) customized to the participant's nutrition-sensitive medical condition(s).
  Interventions: Other: Medically tailored meals
- Medically tailored meals plus enhanced nutritional counseling (Active Comparator): Receive medically-tailored meals only (1 meal per day for total of 10 weeks) with up to 3 remotely delivered enhanced nutritional counseling sessions that are customized to the participant's nutrition-sensitive medical condition(s).
  Interventions: Other: Medically tailored meals
- Usual care (Placebo Comparator): Receive usual standard of care.
  Interventions: Other: Medically tailored meals

INTERVENTIONS:
Other: Medically tailored meals — Compare medically tailored meals vs. medically tailored meals with enhanced nutritional counseling vs. usual care

SUMMARY:
This study is a virtual, remote, decentralized pragmatic clinical trial comparing the efficacy of medically tailored meals alone or medically tailored meals with remote nutritional counseling compared with usual standard of care in adults with a targeted, nutrition-sensitive chronic medical condition (heart failure, diabetes mellitus, chronic kidney disease).

DETAILED DESCRIPTION:
For the KP NOURISH Study, eligible members hospitalized within participating Kaiser Permanente Northern California medical centers will be identified and screened electronically and pre-randomized to 1 of 3 arms (medically tailored meals alone vs. medically tailored meals with remotely delivered enhanced nutritional counseling sessions vs. usual care). Patients enrolled in the medically tailored meals arm will receive 1 medically-tailored meal per day for 10 weeks after hospital discharge. Patients enrolled in the medically tailored meals with enhanced nutritional counseling arm will receive 1 medically-tailored meal per day for 10 weeks after discharge with up to 3 remotely delivered nutritional counseling sessions with a registered dietician nutritionist during the same time period. Patients enrolled in the usual care arm will continue to receive their typical standard of care management. All enrolled patients will complete a questionnaire for patient-reported outcomes (i.e., self-efficacy, social isolation, patient satisfaction, and caring science domains) at baseline and at 10 weeks after discharge and followed electronically for total resource utilization and 30-, 60-, and 90-day outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized at Kaiser Permanente Santa Rosa, Santa Clara, San Francisco, Oakland, or San Rafael Medical Centers
* Kaiser Permanente member at admission
* Has a prior history of at least one of the following:

  1. Heart failure
  2. Diabetes mellitus
  3. Chronic kidney disease

Exclusion Criteria:

* Receiving primary care at Kaiser Permanente facilities outside of Kaiser Permanente Santa Rosa, Santa Clara, San Francisco, Oakland, or San Rafael Medical Centers
* Language interpreter needed
* Admitted from skilled nursing facility or nursing home
* Homeless at admission
* Residence outside the geographic area covered by the medically tailored meals vendors
* Prior history of organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Actual)
Dates: Start 2020-04-27 (Actual); Primary Completion 2021-09-29 (Actual); Study Completion 2021-09-29 (Actual)

PRIMARY OUTCOMES:
90-day hospitalization for any cause | 90-days after discharge from the index hospitalization
  Occurrence of an acute hospitalization for any reasons within 90-days after discharge from the index hospitalization.

SECONDARY OUTCOMES:
90-day hospitalization related to heart failure | 90-days after discharge from the index hospitalization
  Occurrence of hospitalization for heart failure within 90 days after discharge from the index hospitalization.
90-day hospitalization related to diabetes | 90-days after discharge from the index hospitalization
  Occurrence of hospitalization for a diabetes-related complication within 90 days after discharge from the index hospitalization.
90-day all-cause mortality | 90-days after discharge from the index hospitalization
  Occurrence of death from any cause within 90 days after discharge from the index hospitalization.
Patient-reported outcomes | 10 weeks after discharge from the index hospitalization
  Isolation measured on Likert scale (1-5) for 4 different questions related to feelings of isolation. Self-efficacy measured on Likert scale (1-10) for 4 different questions related to feelings of self-efficacy in maintaining healthy dietary habits. Caring science measured on Likert scale (1-5) one question of the impact of meal delivery programs on feelings of being cared for through food.
Emergency department visit for any cause | 30-, 60- and 90-days after discharge from the index hospitalization
  Occurrence of an emergency department visit for any reason within 90 days after discharge from the index hospitalization.
30-day hospitalization for any cause | 30-days after discharge from the index hospitalization
  Occurrence of hospitalization for any reason within 30 days after discharge from the index hospitalization.
60-day hospitalization for any cause | 60-days after discharge from the index hospitalization
  Occurrence of hospitalization for any reason within 60 days after discharge from the index hospitalization.
90-day composite of hospitalization for any cause, emergency department visit for any cause or all-cause death | 90-days after discharge from the index hospitalization
  Occurrence of hospitalization, emergency department visit, or death from any cause within 90 days after discharge from the index hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Alan S Go, MD, Principal Investigator — Kaiser Permanente Northern California Division of Research
Locations (5):
- United States (5):
  - Kaiser Permanente Northern California, Oakland, California
  - Kaiser Permanente Northern California, San Francisco, California
  - Kaiser Permanente Northern California, San Rafael, California
  - Kaiser Permanente Northern California, Santa Clara, California
  - Kaiser Permanente Northern California, Santa Rosa, California

IPD SHARING:
Plan to Share IPD: No